CLINICAL TRIAL: NCT02493699
Title: The Effect of Karate Techniques Training on Communication Deficit of Children With Autism Spectrum Disorders
Brief Title: Martial Arts Therapy in Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Isfahan (Other)
Responsible Party: Principal Investigator, Fatimah Bahrami, Miss, University of Isfahan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/02/2011
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): physical exercise- based intervention (Karate techniques training)
  Interventions: Other: physical exercise- based intervention (Karate techniques training)
- Control (No Intervention): Not participating in physical exercise- based intervention (Karate techniques training)

INTERVENTIONS:
Other: physical exercise- based intervention (Karate techniques training)
  Arms: Exercise

SUMMARY:
The purpose of the present study was to determine whether teaching Karate techniques training leads to reduction in communication deficit of children with autism spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed as autism spectrum disorders according to the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition, Text Revision.
* Age range in 5 to 16.

Exclusion Criteria:

* Not participating in up to 3 intervention sessions.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Raw score of communication subscale of Gilliam Autism Rating Scale-Second Edition (GARS-2) as the measure of communication deficit | within the first 30 days after termination of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fatimah Bahrami, MS, Principal Investigator — University of Isfahan